CLINICAL TRIAL: NCT05615272
Title: A Clinical Investigation of the Efficacy of Platelet Rich Fibrin (Bio-PRF) Compared to Alveogyl in the Treatment of Alveolar Osteitis
Brief Title: Treatment of Alveolar Osteitis: Traditional or Regenerative?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Maeve Cooney, Postgraduate Student in Oral Surgery, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0733
Record Dates: First submitted 2022-10-24; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Alveolar Osteitis; Dry Socket; Pain; Healing; Tooth Extraction
MeSH Terms: conditions — Dry Socket; Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bio-PRF (Experimental): This is a blood-derived platelet rich concentrate from the patient's whole blood sample. The patient typically donates two 9ml (1.5 tablespoons) vials of blood that is then spun in a centrifuge.
  Interventions: Biological: Bio-PRF
- Alveogyl (Active Comparator): Alveogyl is an intraalveolar sedative, obtundent dressing, which contains the active ingredient eugenol.
  Interventions: Drug: Alveogyl

INTERVENTIONS:
Biological: Bio-PRF — Intervention group
  Other Names: Blood Sample
  Arms: Bio-PRF
Drug: Alveogyl — Control group
  Other Names: Intraalveolar Dressing
  Arms: Alveogyl

SUMMARY:
Alveolar osteitis, commonly referred to as dry socket, is a common painful postoperative complication following tooth extraction. It is defined as pain in and around an extraction socket which increases at any time between one and three days following extraction, accompanied by partial or total loss of the blood clot from the socket, with or without halitosis (Blum, 2002).

The incidence of the complication varies from 1-5% for routine extractions up to approximately 30% for third molar extractions. There are a variety of factors that contribute to the incidence of dry socket including tissue trauma, smoking in the early postoperative period and the oral contraceptive pill. Although it is a self- limiting condition, symptoms can be very debilitating for patients and therefore following diagnosis, immediate treatment should be provided to expedite resolution and to their improve quality of life during the healing period. Treatment options for dry socket vary from rinsing of the socket, regular analgesia and sometimes placement of an obtundent, sedative dressing such as Alveogyl or a zinc oxide eugenol alternative.

This study will aim to compare two treatments for patients who present with alveolar osteitis (dry socket) to Dublin Dental University Hospital after tooth extraction. Following randomisation, one of two treatment modalities will be used, either a experimental treatment (Bio-PRF) or a positive control (Alveogyl).

The results of this study will enable us to learn more about the efficacy of these treatment options for dry socket and how they affect patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and females adults at least 18 years old
* A diagnosis of alveolar osteitis following tooth extraction based on patients having both pain and exposed bone
* Good command of the English language
* Willingness to keep a diary of symptoms and travel for the review appointment on day 7 following intervention

Exclusion Criteria:

* Pregnant or breastfeeding women
* Current or previous bisphosphonate used or history of radiotherapy to the jaws
* Allergy or intolerance to study materials
* Lack of capacity to consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain levels: Day 0 to Day 3 | Day 3 following intervention
  Pain will be measured using a pain diary with VAS scale (0-100) at baseline and Day 3. The changes in patient pain levels from baseline will be compared to Day 3 for each group.
Change in postoperative pain levels: Day 0 to Day 7 | Day 7 following intervention
  Pain will be measured using a pain diary with VAS scale (0-100) at baseline and Day 7. The changes in patient pain levels from baseline will be compared to Day 7 for each group.

SECONDARY OUTCOMES:
Healing | Day 7 following intervention
  Healing will be measured clinically by second blinded assessor using a modified version of the Landry Healing Index
Quality of Life Measurements (QoL) | Day 7 following intervention
  The patient's QoL will be assessed using a questionnaire modified from the postoperative symptom severity scale (PoSSe) ranging from 1-5, where 1 correlates to no impact on their quality of life and 5 signifies major impact on their quality of life. Higher scores will mean worse outcome if by Day 7, the patient's QoL scores remain high.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Dr Beattie, Study Director — Specialist Oral Surgeon; John Ed Mr O'Connell, Study Director — Consultant Maxillofacial Surgeon
Locations (1):
- Dublin Dental University Hospital, Dublin, Ireland